CLINICAL TRIAL: NCT03024827
Title: Cannabidiol in Children With Refractory Epileptic Encephalopathy: A Phase 1 Open Label Dose Escalation Study (CARE-E)
Brief Title: Cannabidiol in Children With Refractory Epileptic Encephalopathy
Acronym: CARE-E
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Richard Huntsman, MD, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARE-E-01
Record Dates: First submitted 2016-12-16; First posted 2017-01-19 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Epileptic Encephalopathy
Keywords: Infantile Spasms; Lennox Gastaut Syndrome; Doose Syndrome; Continuous Spike Wave in Sleep; Landau-Kleffner Syndrome; Dravet Syndrome; Malignant Migrating Partial Seizures of Infancy (MMPSI)
MeSH Terms: conditions — Spasms, Infantile; Lennox Gastaut Syndrome; Epilepsies, Myoclonic; Landau-Kleffner Syndrome | interventions — Medical Marijuana

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Cannabis Oil (Experimental): CanniMed® 1:20
  Interventions: Drug: CanniMed® 1:20

INTERVENTIONS:
Drug: CanniMed® 1:20 — A cannabidiol (CBD): tetrahydrocannabinol (Δ9 THC) 20:1 ratio product will be provided as an oil-based suspension.
  Other Names: Medical Cannabis Oil

SUMMARY:
This study will assess the safety and tolerability of a cannabidiol-enriched Cannabis Herbal Extract in a small group of children with refractory epileptic encephalopathy. The dosage of Cannabis Herbal Extract will be gradually increased over a four month time period.

DETAILED DESCRIPTION:
Epileptic Encephalopathies are a group of epilepsies that develop in children. These epilepsies can cause frequent and difficult to control seizures. Because of the ongoing seizures, these epilepsies can also cause cognitive impairment and neurological impairment.

In many children with these Epileptic Encephalopathies, seizures are difficult to control with medical treatment, such as anti-convulsants or non-drug treatments like the ketogenic diet (a high fat, adequate-protein, low-carbohydrate diet). This has resulted in a need to find therapies that are effective and better tolerated for children with epileptic encephalopathies.

There is very limited data regarding the use of cannabis products in children, in particular cannabidiol-enriched cannabis oil in children with epilepsy. However, hemp oil products with high cannabidiol and low tetrahydrocannabinol ratios have been reported to provide seizure relief and cognitive improvement in children who take them.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-10 years
* Epileptic Encephalopathy
* A minimum of at least 1 major seizure per week or 4 major seizures per month. For the purposes of this research study, a major seizure would include atonic, tonic, clonic, tonic-clonic, major myoclonic, myoclonic astatic seizures and epileptic spasms (including infantile spasms)
* Refractory to anticonvulsant medication as per the International League Against Epilepsy (ILAE) Definition of failing 2 appropriate anticonvulsants at therapeutic doses
* The ability to attend appointments regularly
* Negative pregnancy test at screening for females who have reached menarche

Exclusion Criteria:

* Recent (<1 month) change in anticonvulsant therapies including anticonvulsant medications, ketogenic diet or settings on Vagal Nerve Stimulator
* Recent (<6 months) change in intravenous immunoglobulin (IVIG) treatment
* Initiation of ketogenic diet within 6 months (Patients must be on the ketogenic diet for at least 6 months to prevent any delayed response from the ketogenic diet affecting study results)
* Implantation and activation of Vagal Nerve Stimulator within 12 months (Patients may have a vagal nerve stimulator for at least one year once again to prevent delayed response from the vagal nerve stimulator affecting study results)
* Use of cannabis-based therapy within 2 months (Participants who have previously used a cannabis based therapy may be included if they have a 2 month period without use of cannabis based therapy prior to enrolment in the study)
* Use of selective serotonin reuptake inhibitor (SSRI), tricyclic antidepressant or atypical neuroleptic medication in last month
* Concomitant regular use of narcotics (Use of narcotics in emergency situations and supervised by a physician is allowed)
* Initiation or dosage change of oral or injected steroids within 3 months
* Allergy or known intolerance to any of the compounds within the study preparation
* Inability of study participants to attend assessments on a monthly basis
* Clinically significant cardiac, renal or hepatic disease (as assessed by the site investigator)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Up to 6 months
Blood Pressure | Up to 6 months
Weight | Up to 6 months
Complete Blood Count (CBC) and Differential | Up to 6 months
Sodium, potassium, chloride, calcium, magnesium, phosphate and carbon dioxide (mmol/L) | Up to 6 months
Blood Urea Nitrogen (mmol/L) | Up to 6 months
Creatinine (umol/L) | Up to 6 months
Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Gamma-glutamyl transferase (GGT) and Lipase (U/L) | Up to 6 months
Total and Direct Bilirubin (umol/L) | Up to 6 months
Albumin (g/L) | Up to 6 months
Total Cholesterol and Triglyceride (mmol/L) | Up to 6 months
Clobazam and Norclobazam Levels (umol/L) | Up to 6 months
  For participants taking clobazam who become excessively sedated
Clonazepam Level (umol/L) | Up to 6 months
  For participants taking clonazepam who become excessively sedated
Urine Ketones | Up to 6 months
  For participants on the ketogenic diet
Trough Level of Concomitant Anti-Convulsants | Up to 7 months
  Measure interactions with any anti-convulsants participants may be already on
Adverse Events | Through study completion, up to 7 months
  Side effect rating scale, includes items related to sleepiness/lethargy, irritability, nausea/vomiting and diarrhea
2-hour Electroencephalogram (EEG) Recording | Up to 6 months

SECONDARY OUTCOMES:
Seizure Frequency Log Book | Through study completion, up to 7 months
Modified Quality of Life in Children with Epilepsy Questionnaire (QOLCE) | Through study completion, up to 7 months
Cannabidiol (CBD) (ng/mL) | Up to 7 months
  Levels in blood
Tetrahydrocannabinol (Δ9-THC) (ng/mL) | Up to 7 months
  Levels in blood
11-nor-9-carboxy-tetrahydrocannabinol (11-nor-9-Carboxy-THC) (ng/mL) | Up to 7 months
  Levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Richard Huntsman, MD, Principal Investigator — Dalhousie University; Richard Tang-Wai, MD, Principal Investigator — Loma Linda University; Jane Alcorn, PhD, Principal Investigator — University of Saskatchewan
Locations (4):
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Universite de Montreal, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reithmeier D, Tang-Wai R, Seifert B, Lyon AW, Alcorn J, Acton B, Corley S, Prosser-Loose E, Mousseau DD, Lim HJ, Tellez-Zenteno J, Huh L, Leung E, Carmant L, Huntsman RJ. The protocol for the Cannabidiol in children with refractory epileptic encephalopathy (CARE-E) study: a phase 1 dosage escalation study. BMC Pediatr. 2018 Jul 7;18(1):221. doi: 10.1186/s12887-018-1191-y. PMID 29981580
- [Result] Huntsman RJ, Tang-Wai R, Alcorn J, Vuong S, Acton B, Corley S, Laprairie R, Lyon AW, Meier S, Mousseau DD, Newmeyer D, Prosser-Loose E, Seifert B, Tellez-Zenteno J, Huh L, Leung E, Major P. Dosage Related Efficacy and Tolerability of Cannabidiol in Children With Treatment-Resistant Epileptic Encephalopathy: Preliminary Results of the CARE-E Study. Front Neurol. 2019 Jul 3;10:716. doi: 10.3389/fneur.2019.00716. eCollection 2019. PMID 31333569
- See also: Dosage Related Efficacy and Tolerability of Cannabidiol in Children With Treatment-Resistant Epileptic Encephalopathy: Preliminary Results of the CARE-E Study — https://www.frontiersin.org/articles/10.3389/fneur.2019.00716/full